CLINICAL TRIAL: NCT01131923
Title: An Open-Label Randomized Single-Dose Bioequivalence Study of Amlodipine 10 mg Tablets and Norvasc ® 10 mg Tablets Under Fasting Conditions
Brief Title: Bioequivalency Study of Amlodipine Besylate Tablets, 10 mg of Dr. Reddy's Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: M.S. Mohan/Senior Manager R&D, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AAI-US-132
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2010-06-14 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Bioequivalence; Amlodipine Besylate
MeSH Terms: interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amlodipine Tablets, 10 mg (Experimental): Amlodipine Tablets, 10 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Amlodipine
- Norvasc Tablets, 10 mg (Active Comparator)
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Amlodipine — Amlodipine Tablets, 10 mg
  Other Names: Norvasc 10 mg tablets of Pfizer, Inc.,

SUMMARY:
The purpose of this study is to determine the pharmacokinetics and bioequivalence of amlodipine besylate formulations under fasting conditions.

DETAILED DESCRIPTION:
This study evaluates the pharmacokinetics and bioequivalence of Amlodipine Tablets 10 mg of Dr. Reddy's versus Norvasc 10 mg tablets administered as 1 x 10 mg tablet in healthy volunteers with a washout period of 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects between 18 and 45 years of age inclusive.
* Informed of the nature of the study and given written informed consent.
* Have a body weight within 15% of the appropriate range as defined in the 1983 Metropolitan Life Company tables and weigh at least 115 (Appendix I and Appendix II).

Exclusion Criteria:

* If female, the subject is lactating or has a positive pregnancy test at screening and prior to each of the three treatment periods. Females must use a medically acceptable method of contraception throughout the entire study period and for one week after the study is completed. Medically acceptable methods of contraception that may be used by the subject and/or her partner are: oral contraceptives, progestin injection or implants, condom with spermicide, diaphragm with spermicide, IUD, vaginal spermicidal suppository, surgical sterilization of themselves or their partners or abstinence. Females taking oral contraceptives must have taken them consistently for at least three months prior to receiving study medication.
* Hypersensitivity to amlodipine besylate (Norvasc®) or related calcium channel blockers).
* Any history of a clinical condition that might affect drug absorption, metabolism or excretion.
* Recent history of mental illness, drug addiction, drug abuse or alcoholism.
* Donation of greater than 500 ml of blood in the past 4 weeks prior to study dosing or difficulty in donating blood.
* Received an investigational drug within the 4 weeks prior to study dosing.
* Currently taking any prescription medication, except for oral contraceptives, within the 7 days prior to study dosing or over-the-counter medication within 3 days of study dosing. This prohibition does not include vitamins or -herbal preparations taken as nutritional supplements for non-therapeutic indications as judged by the attending physician.
* Regular tobacco use in the 6 months prior to study dosing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2002-10; Primary Completion 2002-11 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Scallion EE, MD, Principal Investigator — AAI Clinic
Locations (1):
- AAI Clinic, Chapel Hill, North Carolina, United States